CLINICAL TRIAL: NCT04711187
Title: A Phase I Study Assessing the Safety and Pharmacokinetics of Multiple Doses of AT-527 in Healthy Subjects
Brief Title: Study of AT-527 in Healthy Subjects (R07496998)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AT-03A-002
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteer Study

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- AT-527 Formulation 1 Dose 1 (Experimental)
  Interventions: Drug: AT-527 Formulation 1; Other: Placebo Comparator
- AT-527 Formulation 2 Dose 1 (Experimental)
  Interventions: Drug: AT-527 Formulation 2
- AT-527 Formulation 2 Dose 2 (Experimental)
  Interventions: Other: Placebo Comparator; Drug: AT-527 Formulation 2
- AT-527 Formulation 1 Dose 3 (Experimental)
  Interventions: Drug: AT-527 Formulation 1; Other: Placebo Comparator
- AT-527 Formulation 2 Dose 3 (Experimental)
  Interventions: Other: Placebo Comparator; Drug: AT-527 Formulation 2
- AT-527 Formulation 2 Dose 1 Fast/Fed (Experimental)
  Interventions: Drug: AT-527 Formulation 2
- AT-527 Formulation 2 Dose 3 Fast/Fed (Experimental)
  Interventions: Drug: AT-527 Formulation 2

INTERVENTIONS:
Drug: AT-527 Formulation 1 — AT-527 Formulation 1 (R07496998)
  Arms: AT-527 Formulation 1 Dose 1; AT-527 Formulation 1 Dose 3
Other: Placebo Comparator — Placebo Comparator
  Arms: AT-527 Formulation 1 Dose 1; AT-527 Formulation 1 Dose 3; AT-527 Formulation 2 Dose 2; AT-527 Formulation 2 Dose 3
Drug: AT-527 Formulation 2 — AT-527 Formulation 2 (R07496998)
  Arms: AT-527 Formulation 2 Dose 1; AT-527 Formulation 2 Dose 1 Fast/Fed; AT-527 Formulation 2 Dose 2; AT-527 Formulation 2 Dose 3; AT-527 Formulation 2 Dose 3 Fast/Fed

SUMMARY:
This study will assess the safety, tolerability and pharmacokinetics (PK) of AT-527 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use two methods of birth control from Screening through 90 days after administration of the last dose of study drug
* Females must have a negative pregnancy test at Screening and prior to dosing
* Minimum body weight of 50 kg and body mass index (BMI) of 18-32 kg/m2
* Willing to comply with the study requirements and to provide written informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Infected with hepatitis B virus, hepatitis C virus, HIV or COVID-19
* Abuse of alcohol or drugs
* Use of other investigational drugs within 28 days of dosing
* Other clinically significant medical conditions or laboratory abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Proportions (active vs. placebo) of subjects experiencing treatment-emergent adverse events. | Day 10

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of AT-527 | Days 1 and 5
  Maximum plasma concentration (Cmax)
Pharmacokinetics (PK) of AT-527 | Days 1 and 5
  Area under the concentration-time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Montreal, Quebec, Canada